CLINICAL TRIAL: NCT02969486
Title: Prospective Proof-of-concept Study Non-invasive Estimation of Pulmonary Artery Pressure in Healthy Subjects by Electrical Impedance Tomography
Brief Title: Non-invasive Estimation of Pulmonary Artery Pressure in Healthy Subjects by Electrical Impedance Tomography
Acronym: PAP-EIT
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00747
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Pulmonary Artery Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Pulmonary hypertension (PH) is a condition characterized by a sustained elevation in pulmonary artery pressure (PAP) above 25 mmHg assessed by right heart catheterization. PH is fatal in absence of adequate treatment or therapy, as the condition progressively increases the workload of the right heart and ultimately leads to its failure. With a minimal indicative prevalence of 1 case/300, PH affects at least 25'000 people in Switzerland alone. After initiation of PH therapy, the follow-up of the patient's health status is often limited to punctual PAP measurements at the clinic at intervals of several months. The lack of more frequent measurements of the patient's PAP strongly hinders the identification of short-term trends in pulmonary hemodynamics, and therefore the anticipation of worsening conditions or treatment inefficiency. As possible solutions, wireless implantable hemodynamic monitors such as the CardioMEMSTM HF System (CardioMEMS Inc., Atlanta, USA) have recently been introduced for the continuous monitoring of PAP in patients with PH. The benefits of frequent measurements over intermittent clinic visits have been demonstrated in several previous studies, notably in terms of prediction of therapy outcomes, anticipation of worsening heart failure, feedback rapidity during therapy, or decline in hospitalization rates. Nevertheless, despite the undeniable advantages that implantable monitors offer to the patient, they remain highly invasive solutions. In contrast, noninvasive alternatives for the measurement of PAP exist, such as transthoracic echocardiography, but are impractical for frequent PAP assessments due to their dependency on qualified personnel to perform the measurement. An optimal PAP monitoring modality for patients with PH should be non-invasive (free of any risks or complications associated with cardiac catheterization) and unsupervised (able to operate without supervision of a medical doctor). Such a modality does not currently exist. In the present study, the investigators propose and investigate the potential of a novel non-invasive, continuous and unsupervised PAP monitoring approach based on the pulse wave velocity (PWV) principle and the use of electrical impedance tomography (EIT).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects ≥ 18 years old, BMI < 30 kg/m2
* Good understanding of written and oral German
* Willing to provide a signed informed consent

Exclusion Criteria:

* Pace-maker/ ICD
* Chronic heart diseases
* Chronic pulmonary diseases
* Congenital heart/pulmonary diseases
* Instable angina pectoris
* Active alcohol or drug abuse
* Pregnancy or lactation (women of childbearing age will be asked to performed urinary pregnancy test before the screening phase)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects ≥ 18 years old
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Correlation coefficients | Single visit 2 hours
  Assessment of significant subject-wise correlation coefficients between the reference PAP, obtained by the gold Standard transthoracic echocardiography technique, and an EIT-derived PAP-related parameter. The primary outcome is therefore the demonstration of the feasibility of monitoring changes in PAP (intra-subject trending ability) by EIT.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Rimoldi, Prof, Study Director — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Background] Strange G, Playford D, Stewart S, Deague JA, Nelson H, Kent A, Gabbay E. Pulmonary hypertension: prevalence and mortality in the Armadale echocardiography cohort. Heart. 2012 Dec;98(24):1805-11. doi: 10.1136/heartjnl-2012-301992. Epub 2012 Jul 3. PMID 22760869
- [Background] McGoon MD, Kane GC. Pulmonary hypertension: diagnosis and management. Mayo Clin Proc. 2009 Feb;84(2):191-207. doi: 10.4065/84.2.191. PMID 19181654
- [Background] Abraham WT, Adamson PB, Bourge RC, Aaron MF, Costanzo MR, Stevenson LW, Strickland W, Neelagaru S, Raval N, Krueger S, Weiner S, Shavelle D, Jeffries B, Yadav JS; CHAMPION Trial Study Group. Wireless pulmonary artery haemodynamic monitoring in chronic heart failure: a randomised controlled trial. Lancet. 2011 Feb 19;377(9766):658-66. doi: 10.1016/S0140-6736(11)60101-3. PMID 21315441